CLINICAL TRIAL: NCT05294887
Title: First Prospective Randomized Trial to Examine a Differential Therapeutic Response in Symptomatic Patients With Non-obstructive Coronary Artery Disease After Coronary Physiological Testing
Brief Title: Randomized Trial to Examine a Differential Therapeutic Response in Symptomatic Patients With Non-obstructive Coronary Artery Disease
Acronym: EXAMINE-CAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Ulf Landmesser, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXAMINE-CAD-DZHK22; 2020-004717-12 (EudraCT Number)
Record Dates: First submitted 2022-02-28; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Coronary Microvascular Dysfunction; Microvascular Angina; Vasospasm, Coronary; Vasospastic Angina; Prinzmetal Angina; Coronary Artery Disease
Keywords: Coronary Microvascular Dysfunction; Microvascular Angina; Coronary Vasospasm; Vasospastic Angina; Beta Blocker; Calcium Channel Blocker
MeSH Terms: conditions — Microvascular Angina; Coronary Vasospasm; Angina Pectoris, Variant; Coronary Artery Disease | interventions — Bisoprolol; Adrenergic beta-Antagonists; Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomly assigned to 1 of 6 possible treatment sequences. All treatment sequences will include the consecutive treatment with bisoprolol, diltiazem, and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- bisoprolol first, diltiazem second (Experimental): Crossover Design: bisoprolol first, diltiazem second, placebo third
  Interventions: Drug: Bisoprolol; Drug: Diltiazem; Drug: Placebo
- bisoprolol first, placebo second (Experimental): Crossover Design: bisoprolol first, placebo second, diltiazem third
  Interventions: Drug: Bisoprolol; Drug: Diltiazem; Drug: Placebo
- diltiazem first, bisoprolol second (Experimental): Crossover Design: diltiazem first, bisoprolol second, placebo third
  Interventions: Drug: Bisoprolol; Drug: Diltiazem; Drug: Placebo
- diltiazem first, placebo second (Experimental): Crossover Design: diltiazem first, placebo second, bisoprolol third
  Interventions: Drug: Bisoprolol; Drug: Diltiazem; Drug: Placebo
- placebo first, bisoprolol second (Experimental): Crossover Design: placebo first, bisoprolol second, diltiazem third
  Interventions: Drug: Bisoprolol; Drug: Diltiazem; Drug: Placebo
- placebo first, diltiazem second (Experimental): Crossover Design: placebo first, diltiazem second, bisoprolol third
  Interventions: Drug: Bisoprolol; Drug: Diltiazem; Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol — beta-adrenergic receptor blocker
  Other Names: beta blocker
Drug: Diltiazem — calcium channel blocker
Drug: Placebo — Placebo

SUMMARY:
EXAMINE-CAD-DZHK22 is a prospective, randomized, double-blind, placebo-controlled, crossover trial investigating the efficacy of beta blocker (bisoprolol) and calcium channel blocker (diltiazem) therapy in symptomatic patients with non-obstructed coronary arteries according to coronary physiological testing results.

DETAILED DESCRIPTION:
Patients presenting with recurrent angina but non-obstructed coronary arteries are increasingly recognized and have a high morbidity and symptomatic burden. These patients are often misdiagnosed and discharged without further investigation or treatment. Current European Society of Cardiology (ESC) guidelines for the management of patients with chronic coronary syndromes recommend beta blockers or calcium channel blockers, depending on the presence of abnormal vasodilatation or abnormal vasoconstriction. Scientific evidence to support this recommendation, however, is scarce and no randomized clinical trial of this differential therapy has been performed in these patients. The aim of the EXAMINE-CAD-DZHK22 trial is therefore to compare for the first time the efficacy of beta blocker (bisoprolol) and calcium channel blocker (diltiazem) therapy in reducing angina symptoms in symptomatic patients with non-obstructed coronary arteries according to coronary physiology testing results. This study is the first to investigate whether coronary physiology testing can guide therapeutic management of these patients depending on whether abnormalities of vasodilatation or vasoconstriction are present. The EXAMINE-CAD-DZHK22 trial will thus fill an important knowledge and evidence gap in the treatment of these highly symptomatic patients, and has the potential to pave the way for future large-scale clinical trials in symptomatic patients with non-obstructed coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years
* Recurrent angina symptoms provoked by exercise and/or repeated attacks of angina at rest (both at least for 4 weeks)
* Absence of flow-limiting coronary artery stenosis (as defined by any coronary artery diameter reduction >50% or fractional flow reserve ≤0.80)
* Left ventricular ejection fraction (LVEF) >50%
* Written informed consent

Exclusion Criteria:

* Pregnancy, planned pregnancy, or breast-feeding
* Female patients of childbearing potential who are unwilling to use a highly effective contraception method during trial participation according to CTFG. In addition, a negative serum or urine pregnancy test must be available prior to randomization.
* Expected life expectancy <1 year
* Contraindications to withholding nitrates, calcium channel blockers, and beta blockers for 48 hours before invasive coronary reactivity testing (e.g. clinical need for rate control in case of permanent atrial fibrillation, recurrent angina symptoms without any possibility to wihthold ongoing medication)
* Known hypersensitivity or contraindication to bisoprolol or diltiazem or any of its excipients.
* Concomitant therapy with systemic drugs that are strong inhibitors of both CYP3A4 and P-gp (azole antimycotics such as ketoconazole and itraconazole or HIV protease inhibitors such as ritonavir)
* Concomitant therapy with drugs that are strong CYP3A4 inducers (e.g. carbamazepine, phenytoin, rifampicin, St. John's wort)
* Bradycardia (<50/min) at time of randomization
* Symptomatic hypotension (<100 mmHg) at time of randomization
* Cardiogenic shock
* Second and third degree atrioventricular block, sick sinus syndrome, sinoatrial block
* Severe valvular heart disease (grade III)
* Any cardiomyopathy including those with preserved left ventricular ejection fraction (LVEF)
* Chronic obstructive pulmonary disease
* Severe bronchial asthma
* Metabolic acidosis at time of randomization
* Renal failure (creatinine >2.0 mg/dL)
* N-terminal pro B-type natriuretic peptide (NT-proBNP) >300 ng/L
* Known significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) which is associated with moderate or severe hepatic impairment (alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥2.0 upper limit of normal (ULN))
* Untreated pheochromocytoma
* Late stage of peripheral arterial disease or Raynaud's syndrome
* Participation in another clinical trial according to AMG or MPG at the time of randomization and the duration of this trial
* Patients who are unwilling to consent to saving and propagation of pseudonymized medical data for study reasons
* Persons who are legally detained in an official institution
* Persons likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of patient's and investigator's knwoledge
* Persons who may dependent on the Sponsor, the Investigator or the trial sites, are not eligible to enter the trial
* Active coronavirus disease 2019 (COVID-19) at time of randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in angina symptom severity as measured by the Seattle Angina Questionnaire (SAQ) summary score from each period specific baseline to the end of this period (week 4) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of angina symptom severity as measured by the SAQ summary score resulting from the SAQ physical limitation scale, SAQ angina frequency scale, and SAQ quality of life scale. The score ranges from 0 to 100, with the lower the score, the higher the symptom severity and limitations.

SECONDARY OUTCOMES:
SAQ angina stability scale | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Individual SAQ domain to evaluate the disease-specific health status with quantification of patients' symptoms of angina. The score ranges from 0 to 100, with the lower the score, the higher the symptom severity and limitations.
SAQ angina frequency scale | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Individual SAQ domain to evaluate the disease-specific health status with quantification of patients' symptoms of angina. The score ranges from 0 to 100, with the lower the score, the higher the symptom severity and limitations.
SAQ treatment satisfaction scale | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Individual SAQ domain to evaluate the disease-specific treatment satisfaction. The score ranges from 0 to 100, with the higher the score, the higher the treatment satisfaction.
SAQ physical limitation scale | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Individual SAQ domain to evaluate the disease-specific health status with quantification of patients' symptoms of angina and the extent to which their angina affects their functioning. The score ranges from 0 to 100, with the lower the score, the higher the symptom severity and limitations.
SAQ quality of life | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Individual SAQ domain to evaluate the disease-specific health status with the extent to which their angina affects their quality of life. The score ranges from 0 to 100, with the higher the score, the higher the quality of life.
Duke Activity Status Index (DASI) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of functional capacity of patients with cardiovascular disease
Rose dyspnea scale | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of patients' dyspnea level with common activities. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea.
Angina diary (Angina episodes per week) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of angina frequency
Angina diary (nitroglycerin use per week)) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of need for nitroglycerine
Quality of Life (Short Form 36 health survey questionnaire) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Evaluation of health-related quality of life
Psychological symptoms as assessed by Patient Health Questionnaire (PHQ-9) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of symptoms for depression in patients with physical illness or physical complaints
Psychological symptoms as assessed by the Hospital Anxiety Depression Scale (HADS)) | from each period specific baseline to the end of this period, i.e. baseline and 4 weeks; 6 weeks and 10 weeks; 12 weeks and 16 weeks
  Assessment of symptoms for depression and anxiety in patients with physical illness or physical complaints
Functional capacity as assessed by bicycle exercise testing | from baseline (visit 1) to the end of each treatment period (4 weeks, 10 weeks, 16 weeks)
  Assessment of functional capacity in bicycle exercise testing (i.e. maximum load capacity in watt)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Landmesser, Prof. Dr., Study Chair — Charité University, Berlin, Germany; Barbara E Stähli, Prof. Dr., Study Chair — Universitätsspital Zürich
Locations (15):
- Germany (13):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité University Medicine Berlin, Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitäres Herz- und Gefäßzentrum UKE Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Deutsches Herzzentrum München des Freistaates Bayern - Klinik an der Technischen Universität München, München
  - Robert-Bosch-Krankenhaus, Stuttgart
- Switzerland (2):
  - Inselspital, Universitätsspital Bern, Bern
  - Universitäres Herzzentrum Zürich, Universitätsspital Zürich, Zurich